CLINICAL TRIAL: NCT00514397
Title: A Phase II Multi-Centre Study of Concomitant and Prolonged Adjuvant Temozolomide With Radiotherapy in Diffuse Pontine Gliomas
Brief Title: Temozolomide and Radiation Therapy in Treating Young Patients With Pontine Glioma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Purpose: Treatment
Other Study IDs: CCLG-CNS-2007-04; CDR0000560114 (Registry Identifier: PDQ (Physician Data Query)); EU-20746; EUDRACT-2007-001768-60
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood brain stem glioma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — motexafin gadolinium; Temozolomide; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: motexafin gadolinium
Drug: temozolomide
Procedure: adjuvant therapy
Procedure: quality-of-life assessment
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving temozolomide together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving temozolomide together with radiation therapy works in treating young patients with pontine glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the time to death in patients with newly diagnosed diffuse pontine gliomas, when treated with the combination of concomitant low-dose oral temozolomide and radiotherapy, followed by up to 12 months of maintenance therapy with extended low-dose temozolomide.
* To assess the quality of life of patients with diffuse pontine gliomas during and after treatment.

Secondary

* To evaluate the time to tumor progression in patients with newly diagnosed diffuse pontine gliomas, when treated with the combination of concomitant low-dose oral temozolomide and radiotherapy, followed by up to 12 months of maintenance therapy with extended low-dose temozolomide.
* To evaluate and document toxicities from the administration of temozolomide combined with radiotherapy and to further study any toxicities associated with the chronic administration of the extended low-dose temozolomide schedule in this population group.
* To document radiological response to the above treatment with MR imaging and, where available, functional imaging.

OUTLINE: This is a multicenter study.

* Chemoradiotherapy: Patients receive oral temozolomide once daily for 6 weeks (7 days per week) with concurrent radiotherapy (5 days per week).

Patients without evidence of disease progression proceed to maintenance therapy beginning at least 4 weeks after completion of radiotherapy.

* Maintenance therapy: Patients receive oral temozolomide daily on days 1-21. Treatment repeats every 4 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed prior to chemoradiotherapy and prior to course 1 of adjuvant temozolomide and prior to every 3 subsequent courses of adjuvant temozolomide.

After completion of study therapy, patients are followed every 8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion criteria:

* Newly diagnosed diffuse intrinsic lesion centered in the pons on MRI

  * No requirement for histological diagnosis
  * Clinical history < 6 months
* Clinical findings must include at least 1 of the 3 following signs of brainstem tumor:

  * Cranial nerve deficit
  * Long tract signs
  * Ataxia

Exclusion criteria:

* Focal lesions of brainstem
* Predominantly exophytic tumors

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Karnofsky performance status (PS) or Lansky PS 60-100% (unless reason for decrease in status is a direct result of neurological involvement of the brainstem glioma)
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 1,000/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Urea and serum creatinine < 1.5 times upper limit of normal (ULN)
* Total and direct bilirubin < 1.5 times ULN
* AST and ALT < 3 times ULN
* Negative pregnancy test within 7 days prior to administration of temozolomide for women of childbearing potential

Exclusion criteria:

* Frequent vomiting and/or medical condition, that could interfere with oral medication intake (e.g., partial bowel obstruction)
* Pregnant or breast-feeding women

PRIOR CONCURRENT THERAPY:

Exclusion criteria:

* Prior chemotherapy or radiotherapy
* Other concurrent investigational drugs
* Other concurrent chemotherapy, immunotherapy, or biologic therapy

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Estimated)
Dates: Start 2008-01

PRIMARY OUTCOMES:
Overall survival
Quality of life including health status, behavior, and the subjective experience using HUI and SDQ methods

SECONDARY OUTCOMES:
Toxicity, steroid usage, and radiological response
Adverse events, including abnormal laboratory parameters, as assessed by CTC criteria

CONTACTS AND LOCATIONS:
Overall Officials: Simon Bailey, MD, Principal Investigator — Sir James Spence Institute of Child Health at Royal Victoria Infirmary
Locations (21):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Bristol Royal Hospital for Children, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - University College Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales